CLINICAL TRIAL: NCT00835523
Title: OHSS Prevention by GnRH-agonist Triggering of Final Oocyte Maturation and Cryoperservation of All Two-pronucleate Oocytes in Women Undergoing Stimulation for IVF With Gonadotrophins and GnRH-analogues: a Prospective, Observational, Multicentric, Clinical Cohort Study
Brief Title: Ovarian Hyperstimulation Syndrome (OHSS) Prevention With Agonist
Status: Completed | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Georg Griesinger, Director of Department of Reproductive Medicine, University Hospital Schleswig-Holstein
Other Study IDs: OHSS 2009
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Ovarian Hyperstimulation Syndrome
Keywords: frozen-thawed embryo replacement; GnRH agonist; GnRH antagonist; ovarian hyperstimulation
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- OHSS risk

SUMMARY:
The aim of the study is to explore the concept of GnRH-agonist triggering in combination with elective cryopreservation of all 2PN oocytes at larger scale in a pragmatic clinical setting. The question asked is: "Does GnRH-agonist triggering and cryopreservation work", in terms of efficacy and safety, when applied to a larger cohort of patients, and by a number of different centres with different clinical routines.

ELIGIBILITY:
Inclusion Criteria:

* Indication for IVF with ICSI
* Age < 40 years
* < 4 failed previous IVF attempts with embryo transfer
* ovarian stimulation with GnRH-antagonist and gonadotrophins
* >20 follicles >11 mm in mean diameter or E2 >4500 pg/ml on the day , on which it was planned to administer hCG
* willing to participate and able to consent
* patient has not previously received GnRH-agonist as a trigger of final oocyte maturation

Exclusion Criteria:

* None

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: IVF patients
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2008-05; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Cumulative ongoing pregnancy rate (10-12 GWs) per patient within 12 months | 12 months after recruitment

SECONDARY OUTCOMES:
ongoing pregnancy rate/frozen-thawed ET | 12 months after recruitment
Ongoing pregnancy rate/first frozen-thawed ET | 12 months after recruitment
time to pregnancy in weeks | 12 months after recruitment
incidence of OHSS III° | 12 months after recruitment
number of cumulus-oocyte-complexes | 12 months after recruitment
fertilization rate (number COCs/number of 2 PN oocytes | 12 months after recruitment
survival rate (number of vital embryos/number of frozen 2 PN oocytes | 12 months after recruitment

CONTACTS AND LOCATIONS:
Overall Officials: Georg Griesinger, PD Dr. med., Study Chair — Department of Obestrics and Gynecology, University Clinic of Schleswig-Holstein, Campus Luebeck
Locations (10):
- Germany (10):
  - IVF-Augsburg, Augsburg
  - Deutsche Klinik Bad Münder, Bad Münder am Deister
  - Department of Obestrics and Gynecology, University Bonn, Bonn
  - Department of Obestrics and Gynecology, University Cologne, Cologne
  - Interdisziplinäres Kinderwunschzentrum, Düsseldorf
  - University Centre for Reproductive Medicine Franken, Erlangen
  - Department of Obestrics and Gynecology, University Clinic of Schleswig-Holstein, Campus Luebeck, Lübeck
  - Department of Obestrics and Gynecology, University Magdeburg, Magdeburg
  - Kinderwunschpraxis, Tübingen
  - Department of Obestrics and Gynecology, University Wuerzburg, Würzburg